CLINICAL TRIAL: NCT02363335
Title: The Role of Phosphodiesterase Inhibitors in Incretin Secretion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 999915074; 15-AG-N074
Record Dates: First submitted 2015-02-13; First posted 2015-02-16 (Estimated); Last update posted 2025-06-12 (Actual); Status verified 2025-06-09

CONDITIONS: Healthy Volunteers
Keywords: GLP-1; Phosphodiesterase Inhibitor; GIP
MeSH Terms: interventions — Roflumilast; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): randomized, double-blind, placebo-controlled cross-over study
  Interventions: Other: Placebo
- Roflumilast (Experimental): randomized, double-blind, placebo-controlled cross-over study
  Interventions: Other: Placebo; Other: Roflumilast
- Roflumilast/Sitaglip (Experimental): randomized, double-blind, placebo-controlled cross-over study
  Interventions: Other: Placebo; Other: Roflumilast/Sitagliptin
- Sitagliptin (Experimental): randomized, double-blind, placebo-controlled cross-over study
  Interventions: Other: Placebo; Other: Sitagliptin

INTERVENTIONS:
Other: Placebo — mixed meal
Other: Roflumilast/Sitagliptin — Both Roflumilast and Sitagliptin together
  Arms: Roflumilast/Sitaglip
Other: Sitagliptin — This is already known to increase GLP-1 & GIP secretion.
  Arms: Sitagliptin
Other: Roflumilast — This is already known to increase GLP-1 & GIP secretion
  Arms: Roflumilast

SUMMARY:
Background:

The drug Roflumilast (Daliresp) is used to treat Chronic Obstructive Pulmonary Disease (COPD). COPD is a lung disease that makes it difficult to breathe. Studies have shown that this drug decreased the blood sugar of people with type 2 diabetes. Sitagliptin (Januvia) is a medication presently used to treat diabetes. Researchers think that both of these drugs may decrease blood sugar by causing an increase in the hormone GLP-1.This hormone is secreted in the small intestines and stomach and is also known as an incretin. Researchers want to study how these drugs affect blood sugar, insulin, and other hormones in the blood.

Objectives:

* To study the effects of Roflumilast (Daliresp) and Sitagliptin (Januvia) on blood sugar and insulin.
* To better understand GLP-1 and other gut hormones. This may lead to new treatments for type 2 diabetes.

Eligibility:

* Healthy volunteers age 21 55.
* Body Mass Index (BMI) less than 30

Design:

-This study will require one screening visit and four study visits, scheduled about 3-weeks apart.

Screening visit requires participants to arrive after fasting for 10 hours and have the following:

* Medical history, physical exam, height, weight, blood pressure measurements and blood and urine tests.
* A 2-hour oral glucose tolerance test (OGTT). Participants will drink an orange-flavored drink containing 75 grams of sugar (300 calories). A blood sample will be taken prior to drinking the beverage and 2-hours later.
* An electrocardiogram (EKG) to measure the electrical activity of the heart.
* Questionnaires about risk for depression or suicide.

Study visits 1to 4:

* Participants will arrive the evening prior and blood work will be done to confirm eligibility. They will not eat or drink anything except water starting at 8:00 p.m.
* About 6:30 a.m. the following day, an I.V. (small plastic tube) will be placed in an arm vein and used to take 20 blood samples over a period of about 11 hours.
* Participants will receive one of the following study medication/placebo groupings in random order:

  1. Roflumilast (Daliresp) 500 mcg pill; and 1 placebo pill
  2. Sitaglipitin (Januvia) 100 mg pill; and 1 placebo pill
  3. Roflumilast (Daliresp) 500 mcg pill; and Sitagliptin (Januvia) 100 mg pill
  4. 2 placebo pills
* One hour later, they will have a 10-hour mixed meal test (MMT). They will be asked to drink a nutritional shake (Ensure Plus). Blood samples will be taken over the next 10 hours to measure blood sugar, insulin and other hormones. At the end of the test, they will be given a meal.
* Participants will answer questions about side effects and symptoms. They will receive a follow-up phone call within 10 days.

DETAILED DESCRIPTION:
Objectives and Specific Aims:

We plan to investigate whether phosphodiesterases are involved in the regulation of glucagon-like peptide-1 (GLP-1) secretion from L cells in humans. We hypothesize that: (1) phosphodiesterase-4D (PDE4D) inhibitor (roflumilast) enhance GLP-1 secretion from L cells; (2) PDE4D inhibitor (roflumilast) and DPP4 inhibitor (sitagliptin) have synergistic effect on increasing the amount of circulating active GLP-1.

Experimental Design and Methods:

Twenty healthy adults, age 21-55, will be recruited for this study. This is a randomized, double-blind, placebo-controlled cross-over study. Each subject will serve as his/her own control and each person will have four different study visits spaced about 3 weeks apart. During each visit, they will receive one of the following medications (oral route) in random order:

1. Roflumilast (Daliresp) 500 mcg + Placebo
2. Sitagliptin (Januvia) 100 mg + Placebo
3. Roflumilast (Daliresp) 500 mcg + Sitagliptin (Januvia) 100 mg
4. Placebo

A 10-hr mixed-meal test will be administered 1 hour after the medications and frequent blood-samplings will be done over 10 hours.

Medical Relevance and Expected Outcome:

Preliminary clinical data have shown that phosphodiesterase inhibitors improved glycemic control in type 2 diabetes, and pre-clinical animal data have shown that phosphodiesterase inhibitors enhanced GLP-1 secretion from L cells. The application of novel, pre-clinical findings to an understanding of human biology and pathobiology is of fundamental and critical importance. This study will give us a better understanding of the regulators of GLP-1 secretion in humans, and this new understanding may lead to new treatments for type 2 diabetes.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 21-55 (Age restriction is used to remove age as a confounding factor because (beta) cells function and insulin resistance tend to deteriorate with age and may affect GLP-1 and GIP levels.
  2. Screening laboratory evaluations with no clinically significant abnormal results (minor deviations from normal lab results will be at the discretion of the principal investigator):

     1. fasting comprehensive metabolic panel
     2. complete blood count with differential and platelet
     3. thyroid function test (TSH)
     4. urine drug screen
     5. Point of care urine pregnancy test (for women who are not surgically sterile)
  3. BMI < 30 (participants with BMI greater than or equal to 30 are excluded because obesity has been associated with attenuation in GLP-1 secretion.
  4. Have had a history of stable weight (maintained weight within +/- 5%) over the past year
  5. Have NOT participated in another clinical trial involving any pharmacologic agents within the past 30 days
  6. Able to complete an inform consent
  7. Agree to not participate in other clinical trials within the study period (at the discretion of the study investigator)

EXCLUSION CRITERIA:

1. FPG greater than or equal to 100 mg/dl or 2-hr OGTT greater than or equal to 140 mg/dL (evidence of glucose intolerance or diabetes)
2. History of anemia, or Hemoglobin < 12.5 mg/dL for men and < 11.5 mg/dL for women during screening visit
3. Weight < 110 pounds (due to blood volume requirement)
4. Evidence of illicit drug use
5. History of substance abuse including marijuana within the past 6 months
6. History of smoking any tobacco products within six months prior to screening
7. Alcohol intake > 30 grams (drink more than 2 beers per day OR equivalent amount of alcohol)
8. History of Human Immunodeficiency Virus (HIV) infection
9. History of active or chronic Hepatitis B and/or C infection
10. History of psychiatric illnesses including major depressive disorder, schizophrenia, bipolar disorder
11. Any lifetime history of suicide attempt
12. History of any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the last year
13. Any suicidal ideation of type 4 or 5 on the C-SSRS during any follow-up visits.
14. Patient Health Questionnaire-9 (PHQ-9) score greater than or equal to 10 during screening visit or any follow-up study visits
15. Generalized Anxiety Disorder-7 (GAD-7) score greater than or equal to 10 during screening visit or any follow-up visits
16. History of pancreatitis
17. History of liver or renal diseases
18. History of gastrointestinal or endocrine disorders
19. History of malignancy (unless P.I. determines that there is no impact of the prior malignancy on study outcomes, i.e. basal cell skin cancer)
20. History of coronary disease or clinically significant abnormalities on electrocardiogram
21. History of seizures or other neurologic diseases
22. History of glucocorticoid use (over one month) or other immunosuppressive agents (any), i.e. Imuran, Neoral, Sandimmune, SangCya, basiliximab (Simulect), daclizumab (Zenapax), muromonab (Orthocolone OKT(3)) prednisone (Deltasone, Orasone) within the past six months
23. Use of proton pump inhibitors (PPI s), i.e. Prilosec, Prevacid, Achiphex, Protonix, Nexium, Zegarid
24. Women who are pregnant or nursing/breast-feeding a child
25. Any medical history that, in the opinion of the investigator(s), may make participation of the subject in the study unsafe

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-02-13; Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
PDE4 inhibitor roflumilast enhances GLP-1 secretion from L cells. | 1-10 hours after ingestion
  GIP & GLP-1 response to a mixed meal.

SECONDARY OUTCOMES:
5.PDE4 inhibitor roflumilast and DPP4 inhibitor sitagliptin have synergistic effect on glucose metabolism involving plasma glucose, insulin, ghrelin, glucagon, pancreatic polypeptide, C-peptide and fibroblast growth factor (FGF) 19, 21, 23. | 1-10 hours after ingestion
  The hormones listed are measured by ELISA
4.PDE4 inhibitor roflumilast has an effect on glucose metabolism involving plasma glucose, insulin, ghrelin, glucagon, pancreatic polypeptide, C-peptide and fibroblast growth factor (FGF) 19, 21, 23. | 1-10 hours after ingestion
  The hormones listed are measured by ELISA
3.PDE4 inhibitor roflumilast and DPP4 inhibitor sitagliptin have synergistic effect on elevating circulating active GIP levels. | 1-10 hours after ingestion
  GIP secretion in response to a mixed meal
2.PDE4 inhibitor roflumilast enhances GIP secretion from K cells. | 1-10 hours after ingestion
  GIP secretion in response to a mixed meal
1.PDE4 inhibitor roflumilast and DPP4 inhibitor sitagliptin have synergistic effect on elevating circulating active GLP-1 levels. | 1-10 hours after ingestion
  GLP-1 secretion in response to mixed meal

CONTACTS AND LOCATIONS:
Overall Officials: Chee W Chia, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
NIA IRP are in discussion and a plan has not been finalized.